CLINICAL TRIAL: NCT03432728
Title: Salivary Antioxidant Capacity of Children With Severe Early Childhood Caries (S-ECC) Before and After Complete Dental Rehabilitation
Brief Title: Salivary Antioxidant Capacity Before and After Complete Dental Rehabilitation
Status: Completed | Type: Observational
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Responsible Party: Principal Investigator, Dr Sharat Pani, Program Director - Pediatric Dentistry, Riyadh Colleges of Dentistry and Pharmacy
Other Study IDs: FPGRP/ /43435005/126
Record Dates: First submitted 2018-01-31; First posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Dental Caries in Children
Keywords: Antioxidant Capacity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- S-ECC: Children in their fifth year of life with severe early childhood caries Children selected will require complete dental rehabilitation under general anesthesia All enrolled children will receive treatment of all dental carious lesions under general anesthesia
  Interventions: Procedure: Dental rehabilitation under general anesthesia
- Control: Children age and sex matched with the S-ECC group who are free of dental caries

INTERVENTIONS:
Procedure: Dental rehabilitation under general anesthesia — Dental treatment of all teeth affected by dental caries in a single visit under general anesthesia
  Groups: S-ECC

SUMMARY:
Salivary samples were obtained from 20 children in their fifth year of life diagnosed S-ECC and 20 age and sex matched controls. Complete dental rehabilitation under general anesthesia was performed for the 20 children with S-ECC, and follow up salivary samples were obtained one week and three months post operatively. The TAC was measured using a commercially available Oxygen Radical Absorbance Antioxidant Assay measurement kit (Zen-Bio ORAC™, AMS Biotechnology, Abington UK).

DETAILED DESCRIPTION:
Background: The association of total salivary antioxidant capacity (TAC) to severe early childhood caries (S-ECC) has been studied in the past. It is not clear if TAC is an indicator of the inflammatory response to the lesion or a marker of the disease.

Aim: This study aimed to measure the salivary TAC levels in children with early childhood caries before and after dental treatment and compare the results to caries free children.

Methodology: Salivary samples were obtained from 20 children in their fifth year of life diagnosed S-ECC and 20 age and gendersex matched controls. Complete dental rehabilitation under general anesthesia was performed for the 20 children with S-ECC, and follow up salivary samples were obtained one week and three months post operatively. The TAC was measured using a commercially available Oxygen Radical Absorbance Antioxidant Assay measurement kit (Zen-Bio ORAC™, AMS Biotechnology, Abington UK).

ELIGIBILITY:
Inclusion Criteria:

* Medically fit children
* Age below 71 months
* Test group - to be diagnosed with severe ECC
* Control group - to be caries free

Exclusion Criteria:

Ages: 60 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: * Children who are on long term medications,
  * Children with chronic diseases
  * Children who have had an infection less than three weeks prior to collection of saliva
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2017-01-28 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change in TAC after one week | One week
  Change in Total Salivary Antioxidant Capacity of children from baseline to one week after treatment
Change in TAC after Three months | Three months
  Change in Total Salivary Antioxidant Capacity of children from baseline to three months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sharat C Pani, MDS, Principal Investigator — Riyadh Colleges of Dentistry and Pharmacy
Locations (1):
- Riyadh Colleges of Dentistry and Pharmacy, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No